CLINICAL TRIAL: NCT01445977
Title: SoundBite Hearing System Long Term Multi Site Patient Use Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sonitus Medical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN006
Record Dates: First submitted 2011-09-28; First posted 2011-10-04 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Single Sided Deafness; Conductive Hearing Loss
Keywords: Sonitus Medical; SoundBite; Single Sided Deafness; Conductive Hearing Loss; Unilateral Hearing Loss
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Unilateral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This study is designed to collect data about the SoundBite™ Hearing System to answer specific questions. The hearing system has been cleared for commercial distribution by the Food and Drug Administration (FDA). Sonitus hopes to learn from a larger group of users what features and settings of this device provide the best hearing ability for people diagnosed with Single Sided Deafness (SSD) or Conductive Hearing Loss (CHL).

DETAILED DESCRIPTION:
The Sonitus SoundBite Hearing System prosthetic device is a bone conduction device that has been FDA cleared for treatment of single-sided deafness (SSD) and conductive hearing loss (CHL). The Sonitus SoundBite Hearing System consists of an In the Mouth (ITM) component an external microphone component, worn behind the ear (BTE), a calibration interface cable and PC-controlled calibration software for subject calibration. A charger is also provided to charge the ITM and the BTE. The objective of this multi-sites observational study is to assess the long-term patient use of the Sonitus SoundBite Hearing System.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or older
* Clinical diagnosis of a Moderately severe, severe, or profound sensorineural hearing loss in one ear and normal hearing in the other ear (Normal hearing is defined as a pure tone average (PTA) air-conduction (AC) hearing threshold (measured at 0.5, 1, 2, and 3 kHz) of better than or equal to 25 dB HL)
* Patients diagnosed with conductive hearing loss where the pure tone average bone-conduction hearing threshold (measured at 0.5, 1, 2, and 3 kHz) is better than or equal to 25 dB HL.
* At least two contiguous molar or premolar teeth with no untreated tooth decay. -Patients with tooth decay present are to first have restorations before being fitted for SoundBite
* Healthy attachment to those teeth with tooth pockets limited to no more than 5mm
* No mobile teeth
* Bone loss no greater than a 34% average on the mesial and distal sides of the tooth as measured on X-ray on the teeth on which the device will be worn.

Exclusion Criteria:

* The SoundBite Hearing System and all portions of it are contraindicated for use in an MRI Environment and should be removed prior to MRI exposure
* The SoundBite Hearing System is not to be used in patients with known hypersensitivity to any of the components including allergies to polymers.
* The SoundBite Hearing system is contraindicated for vulnerable populations that are unable to sue their hands such as paraplegics or others that are unable to comply with the warnings in the product's labeling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All trial subjects are individuals that have decided to purchase SoundBite Hearing System for treatment of their Single Sided Deafness or Conductive Hearing Loss and are willing to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Aided Threshold Testing | 12 months
  Aided threshold testing of the impaired ear at 12 months as compared with baseline using the SoundBite Hearing System
Abbreviated Profile of Hearing Aid Benefit (APHAB) Questionnaire | 12 months
  Change in Abbreviated Profile of Hearing Aid Benefit (APHAB, Form A - New Format, Hearing Aid Research Lab, University of Memphis, 1994) score at 12 months compared to baseline
Single Sided Deafness Questionnaire | 12 months
  This questionnaire assesses qualitative outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Popelka, PhD, Principal Investigator — Stanford University
Locations (13):
- United States (13):
  - Arizona Ear Center, Phoenix, Arizona
  - California Hearing and Balance Center, La Jolla, California
  - Shohet Ear Associates Medical Group, Newport Beach, California
  - Camino Ear, Nose and Throat Clinic, San Jose, California
  - Hearing Resource Center, San Mateo, California
  - The George Washington University- Department of Otolaryngology, Washington D.C., District of Columbia
  - University of Miami, Miller School of Medicine, Miami, Florida
  - Physicians Choice Hearing and Dizziness Center, Tampa, Florida
  - Henry Ford Health System- Department of Otolayrngology and Audiology, Detroit, Michigan
  - New York Otology, New York, New York
  - Carolina Ear and Hearing Clinic, PC, Raleigh, North Carolina
  - Ear Medical Group, San Antonio, Texas
  - University Health Science Center (University of Utah Hospital), Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://soundbitehearing.com